CLINICAL TRIAL: NCT03957460
Title: Accuracy of Continuous and Non-invasive Hemoglobin Monitoring During Laparoscopic Gastrectomy: Observational Study
Brief Title: Accuracy of Continuous and Non-invasive Hemoglobin Monitoring
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-17-216
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- continuous and noninvasive hemoglobin monitoring: Group receive the continuous and noninvasive hemoglobin monitoring during laparoscopic gastrectomy.
  Interventions: Other: SpHb monitoring

INTERVENTIONS:
Other: SpHb monitoring — Subjects receive the continuous and noninvasive hemoglobin monitoring (SpHb monitoring).

SUMMARY:
The primary purpose of this observational study is to investigate the accuracy on the continuous and non-invasive hemoglobin monitoring during laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic gastrectomy under general anesthesia

Exclusion Criteria:

* atypical hemoglobin disease, infective state, cardiovascular disease, peripheral vascular disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were scheduled for laparoscopic gastrectomy and recieved the SpHb monitoring during surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
difference between SpHb value in g/dL and SaHb value in g/dL (SpHb - SaHb) | from the start of anesthesia to the end of anesthesia, an average 2 hours
  SpHb value in g/dL is measured by co-oxymetry, and SaHb value in g/dL is measured by blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, South Korea